CLINICAL TRIAL: NCT06746597
Title: Evaluating Mechanical Properties Change Using Optical Coherence Tomography on Plantar Skin Layers
Brief Title: Evaluating Skin Changes Using Optical Coherence Tomography on Plantar Layers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CRREC-112-130
Record Dates: First submitted 2024-12-09; First posted 2024-12-24 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Skin Thickness; Skin Stiffness
Keywords: OCT; skin thickness; skin stiffness; walking intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Three different air-insole presures (80 mmHg, 160 mmHg, and 240 mmHg) (Active Comparator)
  Interventions: Other: Walking intervention on plantar skin thickness and stiffness
- Two different durations (10 and 20 minutes) (Active Comparator)
  Interventions: Other: Walking intervention on plantar skin thickness and stiffness

INTERVENTIONS:
Other: Walking intervention on plantar skin thickness and stiffness — Walking intervention in three different air-insole pressures (80 mmHg, 160 mmHg, 240 mmHg) in two different walking durations (10 and 20 minutes).

SUMMARY:
The goal of this clinical trial is to learn if there are changes in plantar skin surface walking intervention in different air-insole pressures and durations. The main questions it aims to answer are:

How far does walking intervention affect the changes in epidermis layers? What conditions affect the most in the plantar surface, the different air-insole pressures or the different durations?

Researchers will compare the use of three different air-insole pressures (80 mmHg, 160 mmHg, and 240 mmHg) in two different durations (10 and 20 minutes) to see how far the plantar skin surface changes in thickness and stiffness.

Participants will:

Get their plantar region checked and measured by Optical coherence tomography in thickness and stiffness before the walking intervention.

Walk with a custom-made shoe using adjusted air-insole pressures (80 mmHg, 160 mmHg, and 240 mmHg) in two different durations (10 and 20 minutes) Get their plantar region checked and measured by Optical coherence tomography in thickness and stiffness after the walking intervention.

ELIGIBILITY:
Inclusion Criteria:

* Right leg dominant
* Can walk without help

Exclusion Criteria:

* Active ulcers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Measurements of the Stratum Corneum and Deeper Epidermis are recorded in micrometers (for thickness) by comparing baseline values before walking to those obtained after the intervention. | Through study completion, an average of 1 year
  The study involves six walking conditions, each combining one of three air-insole pressures (80 mmHg, 160 mmHg, and 240 mmHg) with either a 10- or 20-minute duration. Each participant completes two conditions daily with a mandatory rest of at least 20 minutes between sessions. Participants can complete all conditions for at least three days by doing two sessions daily or six days with one session per day. This structured approach ensures consistent data collection while minimizing participant fatigue.
  The stratum corneum thickness is measured from the top layer of the stratum corneum to the lower border of the stratum corneum. The deeper epidermis is measured from the lower border of the stratum corneum until the lower border between the epidermis and dermis.

SECONDARY OUTCOMES:
Measurements of the Stratum Corneum and Deeper Epidermis are recorded in megapascal (MPa) or kilopascal (kPa) units (for stiffness) by comparing baseline values before walking to those obtained after the intervention. | Through study completion, an average of 1 year
  The study involves six walking conditions, each combining one of three air-insole pressures (80 mmHg, 160 mmHg, and 240 mmHg) with either a 10- or 20-minute duration. Each participant completes two conditions daily with a mandatory rest of at least 20 minutes between sessions. Participants can complete all conditions for at least three days by doing two sessions daily or six days with one session per day. This structured approach ensures consistent data collection while minimizing participant fatigue.
  The epidermis stiffness is measured by analyzing the changes on the skin after receiving negative pressure suction in 30 kPa from the OCT device.

CONTACTS AND LOCATIONS:
Locations (1):
- Asia University, Taichung, Wufeng, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://drc.bmj.com/content/8/1/e001479
- See also: Related Info — https://journals.lww.com/md-journal/fulltext/2023/10270/the_effects_of_different_inner_pressures_of_air.12.aspx